CLINICAL TRIAL: NCT05752578
Title: Influence of Hot and Cold Cognition on Prospective Memory in HIV+ Patients
Brief Title: Perspective Memory and Executive Functions in HIV+ Patients
Acronym: (3514)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 3514
Record Dates: First submitted 2023-01-30; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with HIV infection: Both male and female subjects, over 18 years of age, on antiretroviral therapy, native speakers of Italian
  Interventions: Other: Neuropsychological testing
- Healthy control subjects: Both male and female subjects, over the age of 18 years, no neurological or psychiatric conditions that would alter test performance, native speakers of Italian
  Interventions: Other: Neuropsychological testing

INTERVENTIONS:
Other: Neuropsychological testing — During the session the patient will be administered the Memory for Intentions Screening Test (MIST; Raskin et al., 2010) with the purpose of investigating prospective memory ability. Then during the same meeting the following tests will be offered to the patient: Montreal Cognitive Assessment (MOCA; Nasreddine. Translation Pirani et al 2006) investigating global cognitive performance; - Interpersonal Reactivity Index (IRI; Davis, 1980;1983- Italian version edited by Bonino et al, 1998) with the purpose of assessing cognitive and affective empathy (Hot cognition); Modified Five Point Test (Ruffi et al 1987) aimed at assessing figurative fluency (Cold cognition).

SUMMARY:
The primary goal of this observational study is to evaluate prospective memory in HIV+ patients compared to healthy subjects. The secondary goal is to examine the relationship between prospective memory and Hot Cognition (mechanical cognitive abilities) and Cold Cognition (cognitive abilities supported by emotion and social perception). The main questions it aims to answer are:

* Do HIV+ patients have more impaired prospective memory than healthy subjects?
* Is there a greater influence of Hot Cognition on prospective memory than Cold Cognition? Participants will undergo a battery of neuropsychological tests: Memory for Intentions Screening Test (MIST), Montreal Cognitive Assessment (MOCA), Interpersonal Reactivity Index and Modified Five Point Test.

ELIGIBILITY:
Inclusion Criteria HIV+:

* consent to participate in the study
* diagnosis of HIV
* Current antiretroviral therapy
* age >18 years
* native Italian speaker

Exclusion Criteria HIV+:

* age <18 years
* presence of major psychiatric disorders within the past 6 months
* additional neurological conditions that may impair the performance of the tests (Alzheimer's disease, Outcomes of head-brain trauma, cerebrovascular episodes)
* Alcohol and drug addiction within the past 6 months
* Additional medical conditions that may impair neurocognitive profile and functional abilities (cerebrovascular damage, cardiac problems with functional impairment, severe liver disease)

Inclusion Criteria HIV- :

* consent to participate in the study
* Absence of HIV infection (HIV-RNA negative)
* age >18 years
* native speaker of Italian

Exclusion Criteria HIV+ :

* age <18 years
* presence of major psychiatric disorders within the past 6 months
* additional neurological conditions that may impair the performance of the tests (Alzheimer's disease, Outcomes of head-brain trauma, cerebrovascular episodes)
* Alcohol and drug addiction within the past 6 months
* additional medical conditions that may impair neurocognitive profile and functional abilities (cerebrovascular damage, heart problems with functional impairment, severe liver disease).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We expect the population with HIV and the healthy population compared by age (between 40 and 60 years old for the majority) and schooling (majority high school graduates). We expect a virologically suppressed HIV population with good adherence to antiretroviral therapy and deficits in prospective memory compared with the healthy population.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Prospective memory in HIV+ patients and healthy subjects | 1 year
  Prospective memory will be assessed through the following test: Memory for Intentions Screening Test (MIST).

SECONDARY OUTCOMES:
Influence of global cognitive performance on prospective memory | 1 year
  Montreal Cognitive Assessment (MOCA) investigating global cognitive performance.
Influence of hot cognition on perspective memory | 1 year
  Interpersonal Reactivity Index (IRI) with the purpose of assessing cognitive and affective empathy (Hot cognition).
Influence of cold cognition on perspective memory | 1 year
  Modified Five Point Test aimed at assessing figurative fluency (Cold cognition).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No